CLINICAL TRIAL: NCT02469987
Title: A Single Center, Randomized, Double-blind, 3-arm Parallel Phase1 Study to Assess PK, Safety, and Tolerability of a Single 90 Min iv Infusion of 1 mg/kg MYL-1402O, EU Avastin®, and US Avastin® in Healthy Male Volunteers
Brief Title: Phase I - Pharmacokinetic Comparability Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MYL-1402O-1002; 2014-005621-12 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: safety; tolerability; immunogenicity; MYL-1402O; PK; Avastin®; biosimilarity; male
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MYL-1402O (Experimental): MYL-1402O (bevacizumab), single 1mg/kg i.v. infusion over 90 minutes.
  Interventions: Drug: MYL-1402O
- US Marketed Avastin (R) (Active Comparator): US Marketed Avastin(R) (bevacizumab), single 1mg/kg i.v. infusion over 90 minutes.
  Interventions: Drug: US marketed Avastin(R)
- EU Marketed Avastin(R) (Active Comparator): EU Marketed Avastin(R) (bevacizumab), single 1mg/kg i.v. infusion over 90 minutes.
  Interventions: Drug: EU marketed Avastin(R)

INTERVENTIONS:
Drug: MYL-1402O — Treatment A - single 1mg/kg dose of MYL-14020 IV infusion over 90 mins.
  Other Names: Bevacizumab
  Arms: MYL-1402O
Drug: US marketed Avastin(R) — Treatment B - single 1mg/kg dose of US marketed Avastin® IV infusion over 90mins
  Other Names: Bevacizumab
  Arms: US Marketed Avastin (R)
Drug: EU marketed Avastin(R) — Treatment C - single 1mg/kg dose of EU marketed Avastin® IV infusion over 90mins.
  Other Names: Bevacizumab
  Arms: EU Marketed Avastin(R)

SUMMARY:
Double-blind, single-dose, three-treatment, parallel group design PK comparability study of MYL-1402O solution manufactured for Mylan compared to US and EU marketed Avastin® solution (bevacizumab).

DETAILED DESCRIPTION:
Double-blind, single-dose, three-treatment, parallel group design PK comparability study of MYL-1402O solution manufactured for Mylan compared to US and EU marketed Avastin® solution (bevacizumab) in a total of 111 healthy, adult male volunteers (37 subjects per treatment arm). After randomization, subjects will receive one of the following treatments: A single 1 mg/kg dose administered by i.v. infusion (25 mL over approximately 90 minutes) of MYL-1402O, an equivalent i.v. infusion of US marketed Avastin® (1 mg/kg), or an equivalent i.v. infusion of EU marketed Avastin® (1 mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-55 yrs. (inclusive)
* BMI: 19.0 to 30.0 kg/m2 (inclusive)
* Weight: ≥ 60kg and ≤100kg
* Subjects should be willing to use adequate contraception and not donate sperm from admission to clinical research center until 6 months post dosing.
* All intermittent medications should have be stopped at least 14days prior to admission to the clinical research center.
* All intermittent non topical medication must be stopped at least 30days prior to admission to the clinical research center.
* Ability and willingness to abstain from ETOH 48hrs prior to admission to the clinical research center.
* Medical history without significant findings per the PI
* Resting supine systolic BP of ≤140mmHg and diastolic BP of ≤90mmHg
* ECGs (via 12 lead) showing NCS findings per PI
* All clinical laboratory tests of blood and urine, WNL and/or without clinically significant findings
* Willing/able to sign ICF
* Normal bowel habits
* Negative medical history regarding fecal blood positivity
* Normal and/or NCS spot protein/creatinine (PCR) ratio.

Exclusion Criteria:

* Previous participation in the current study
* History of prior exposure to bevacizumab
* Evidence of clinically significant findings
* Cognitive and / or mentally impaired handicaps that would affect ability to make an informed consent and/or remain compliant to the requirements of this trial.
* History of relevant drug and/or food related allergies.
* History of or known hypersensitivity to bevacizumab or other recombinant human or humanized antibodies or inactive ingredients.
* Tobacco product use w/I 1 yr. prior to drug administration.
* History of ETOH and or drug abuse/addiction
* Positive urine drug and ETOH screen for opiates, methadone, cocaine, amphetamines including XTC, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and ETOH.
* Average intake of more than 24 units of ETOH / wk. (1 unit of ETOH equals ~250mL of beer, 100mL of wine or 35mL of spirits).
* Consumption of any foods containing poppy seeds w/I 48 hrs. prior to screening and admission to the clinical research center
* Positive screen for Hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies.
* Participation in a drug study w/I 60days or 5 half-lives of the previous drug.
* Participation in more than 3 other drug studies in the 10months prior to drug administration in the current protocol.
* Donation or loss of more than 100mL of blood w/I 60days prior to drug administration. Donation or loss of more than 1.5liters of blood w/I the 10months prior to drug administration.
* Strenuous exercise w/I 96 hrs. Prior to admission to the clinical research center.
* Significant or acute illness w/I 5days prior to drug administration that may impact safety assessments per the judgement of the PI.
* Unsuitable veins for infusion and/or venepuncture
* Surgery including surgery with suturing via a dental procedure or would dehiscence w/I 28days of dosing. Any planned surgery or dental procedures during the study and for at least 30days after follow up.
* Presence of a non-healing wound or fracture.
* History of bleeding disorders
* History of thromboembolic conditions
* History of gastrointestinal perforations or any fistulae.
* History of orthostatic hypotension, fainting spells, blackouts for any reasons.
* History of hypertension
* Medically significant dental disease or dental neglect with signs and or symptoms of local or systemic infection that would likely require a dental procedure during the course of study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for bevacizumab. | pre-dose and 0.33, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, and 2352 hours after start of infusion.
  Area under the plasma concentration versus time curve (AUC) for bevacizumab

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for bevacizumab | pre-dose and 0.33, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 264, 336, 504, 672, 1008, 1344, 1680, 2016, and 2352 hours after start of infusion.
  Area under the plasma concentration versus time curve (AUC) for bevacizumab

OTHER OUTCOMES:
Number of Participants with Adverse Events | up to 99 days.
  Number of Participants with Adverse Events
Safety variable - immunogenicity | Predose day 1, and days 15, 43, 71, and 99 post infusion
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A. Hummel, PhD, Study Director — Mylan Pharmaceuitcals Inc.
Locations (1):
- PRA Health Sciences - Early Development Services, Zuidlaren, Netherlands

REFERENCES:
- [Derived] Hummel M, Bosje T, Shaw A, Liu MS, Barve A, Kothekar M, Socinski MA, Waller CF. A pharmacokinetics study of proposed bevacizumab biosimilar MYL-1402O vs EU-bevacizumab and US-bevacizumab. J Cancer Res Clin Oncol. 2022 Feb;148(2):487-496. doi: 10.1007/s00432-021-03628-0. Epub 2021 Apr 17. PMID 33866430